CLINICAL TRIAL: NCT07377331
Title: Exploration of Structure Retrieval Practice to Support Caregivers' Knowledge Transfer
Brief Title: Exploration of an Online Education Program to Support Caregivers' Knowledge Transfer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Uma Tauber, Professor of Psychology, Texas Christian University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-153-4
Record Dates: First submitted 2026-01-14; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Dementia
Keywords: dementia; caregiving; knowledge; transfer; behaviorial problems
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Longitudinal, behavioral intervention, randomized controlled trial with crossover assignment to condition (SRP vs. Active Control Comparison). Individual-level random assignment will occur for order of the conditions.
Masking Description: Single-blind (outcome assessors blinded to condition assignment). Participants will be masked to study hypotheses, but may detect differences between the SRP and active control conditions during the learning phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within-participant design with 2 learning conditions: intervention and reading control (Experimental): For each caregiver participant, half of the BPSD categories (i.e., 4) will be randomly assigned to the structured retrieval practice (SRP) intervention, and the other half will be randomly assigned to the restudy control condition.
  Interventions: Behavioral: Structured Retrieval Practice (SRP)

INTERVENTIONS:
Behavioral: Structured Retrieval Practice (SRP) — Participants will complete self-paced practice tests for the 4 categories assigned to the SRP intervention. Specifically, the practice test will consist of 24 total questions: 6 multiple-choice questions for each of the 4-categories - 3 questions on triggers and 3 questions on symptom management. Each question will have 1 correct answer and 3 incorrect lures. The vertical order of responses on the screen will be randomized per participant. Questions will be presented in a blocked fashion such that participants will answer all 6 questions in one category (e.g., anxiety), in a random order, before moving to the next (e.g., hallucinations). After each multiple-choice answer, participants will receive detailed, corrective feedback. They will self-pace their study of feedback. Participants will complete 3 practice retrieval blocks.

SUMMARY:
The overarching goal of this work is to determine methods that improve caregiver education about the behavioral and psychological symptoms (BPSD) of dementia. The specific goal of this project is to extend our prior work to evaluate the impact of our educational intervention on caregivers' ability to transfer knowledge about the management of ADRD to real-world applied examples.

ELIGIBILITY:
Inclusion Criteria:

* informal caregivers
* 18+ years old
* Read and speak English
* free of cognitive impairments that prevent consent and/or completing experimental tasks
* remote participants need access to a tablet, laptop, or desktop computer to complete tasks.

Exclusion Criteria:

* professional caregivers
* former caregivers who are not currently caring for someone living with dementia
* caregivers providing assistance to someone with normal cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Immediate near transfer test performance | 10 minutes post-intervention (session 1)
  proportion correct on the immediate (approx. 10 min retention interval) test of near transfer. The test will include 48 questions and will be fill-in-the-blank format. Performance will be explored via percent correct on the test and magnitude of the retrieval practice effect on the test.
immediate applied transfer test performance | approx. 10 minutes post-intervention (session 1)
  proportion correct on the immediate (approx. 10 min retention interval) test to apply examples of symptoms of ADRD. The test will include 8 questions and be short-answer format. Performance will be explored via percent correct on the test and magnitude of the retrieval practice effect on the test.
Delayed Near Transfer test performance | 2 days post-intervention (session 2)
  proportion correct on the final 2-day delayed test of near transfer. The test will include 48 questions and will be fill-in-the-blank format. Performance will be explored via percent correct on the test, magnitude of the retrieval practice effect on the test, and amount of forgetting.
Delayed Applied Transfer test performance | 2 days post-intervention (session 2)
  proportion correct on the final 2-day delayed test of transfer to apply examples of symptoms of ADRD. The test will include 8 questions and be short-answer format. Performance will be explored via percent correct on the test, magnitude of the retrieval practice effect on the test, and amount of forgetting.

SECONDARY OUTCOMES:
Delayed knowledge test performance | 2 days post-intervention (session 2)
  proportion correct on the final 2-day delayed test of symptoms of ADRD. The test will include 48 questions and will be in multiple-choice format. Performance will be explored via percent correct on the test, magnitude of the retrieval practice effect on the test, and amount of forgetting.
Immediate knowledge test performance | 10 minutes post-intervention (session 1)
  proportion correct on the immediate (approx. 10 min retention interval) test of symptoms of ADRD. The test will include 48 questions and will be in multiple-choice format. Performance will be explored via percent correct on the test, magnitude of the retrieval practice effect on the test, and amount of forgetting.
Medical Health Knowledge | 2 days post-intervention (session 2)
  Participants will complete the Medical Term Recognition Test (METER, Rawson et al., 2010). The METER is completed on paper. A list of 40 medical words and 40 nonwords are presented. Participants read the list of items and select the ones that they recognize as real words. Participants are instructed not to guess and to only select items they are sure were real words. Performance on the METER is calculated as the number of words correctly recognized.
Demographic Characteristics | Baseline and 2 days later
  age, gender, education level, race/ethnicity, first generation status, member of an underrepresented group, native language, socioeconomic status, occupation, zip code, relationship with individual living with Alzheimer's Disease or a related dementia (e.g., child, spouse), caregiving status and duration of caregiving, and information seeking about dementia and caregiving.
Self-reported Subjective health information | Baseline and 2 days later
  Caregivers will self-report co-morbid medical conditions for the PLwD, and will report medication use, rating of health, hospitalizations, access to health insurance for the PLwD. Caregivers will be allowed to skip any questions they desire should they prefer not to report responses to any of these questions. No measurement scale will be used for these self-report questions. Instead, these brief questions are intended to obtain general health information. Example questions include, "does the person have other chronic conditions?" "Does the person living with dementia take any prescription medications?" and "Have you gone to the hospital emergency room (ER) about the person living with dementia's health in the past year (12 months)?" Responses to these questions will be used for descriptive purposes to better understand the sample and will not be aggregated into one measure.
Symptom Presence, Severity, and Frequency | pre-intervention, measure occurs online during participant screening
  The behavioral and psychological symptoms experienced by the person living with dementia will be rated by the caregiver participants using the updated version of the Neuropsychiatric Inventory Questionnaire (NPI-Q; Cummings et al., 1994; Resnick et al., 2024; Resnick et al., 2021). This measure includes 12 items that the participant will rate on presence (yes vs. no), severity (1 = mild, 2 = moderate, 3 = severe), and distress (1 = not distressing at all to 5 = extremely distressing). Perceived symptom severity will be measured twice applying a pre-test post-test design.
Performance During Learning | Baseline
  Caregivers' performance during learning will be defined as the percent correct on retrieval practice trials. Specifically, caregivers will respond to multiple choice questions during learning when engaging in retrieval practice, and learning progress will be quantified by aggregating responses across items for each block. Each multiple choice question will have 1 correct answer and 3 incorrect lures, and responses will be scored as 1 (correct) or 0 (incorrect) and then aggregated per participant. This is a quantitative measure that is standard in the science of learning and for which no validated scale is available. Performance on retrieval practice trials for the will be evaluated with item-level analysis (to explore content difficulty) and across each learning block to establish participants' rate-of-learning.
Raven's Progressive Matrices | immediately following intervention during session 1
  Non-verbal fluid intelligence will be assessed with a computerized version of Raven's progressive matrices (Raven, et al., 1998). Participants will complete 18 trials in ascending order in trial normative difficulty (Ariel, Babineau, & Tauber, 2023; adapted from Stanovich & Cunningham, 1993). For each trial, a 3 x 3 array will be displayed with 8 geometric figures. The 9th position in the bottom right-hand corner will be empty. Participants will be given 8 geometric figures from which to choose to correctly complete the array. Participants will be given 10 minutes to complete as many trials as possible. Performance will be calculated as the total number of trials correct.

OTHER OUTCOMES:
Verification of Alzheimer's Disease or Related Dementia (ADRD) | participant screening, pre-intervention
  Verification of ADRD symptoms for each caregiver's person living with dementia (PLwD) is critical to confirm authentic caregiving. We will use the Ascertain Dementia 8 (AD8; Galvin et al., 2005), a validated informant interview sensitive to early cognitive change with strong predictive accuracy (AUC = .83), diagnostic accuracy (AUC = .92; Chen et al., 2018), and cross-cultural validation (Dominguez et al., 2021; Ismail et al., 2021; Meguro et al., 2015). The 3-minute interview will be conducted in-person or via video call. Caregivers answer 8 questions (e.g., Has there been a change in the last several years caused by cognitive (thinking and memory) problems? Have there been problems with judgments (e.g., falls for scams, bad financial decisions, buys gifts inappropriate for recipients) in the last several years?) by responding, yes, no, or N/A (don't know). Scores (0-8) sum affirmative responses; higher scores indicate more impairment. A cutoff ≥ 2 indicates high probability of carin

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Texas Christian University, Fort Worth, Texas
  - Virginia Wesleyan University, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code